CLINICAL TRIAL: NCT01619280
Title: A Phase 1 Study: The Determination of the Maximum Tolerable Dosage of Nebulized Sodium Nitroprusside in Adult Acute Lung Injury
Brief Title: Safety Study of Nebulized Sodium Nitroprusside in Adult Acute Lung Injury
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-0102-A
Record Dates: First submitted 2012-05-29; First posted 2012-06-14 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome; Sodium Nitroprusside; Hypoxia; Respiratory Failure
Keywords: Acute Lung Injury; Acute Respiratory Distress Syndrome; Sodium Nitroprusside; adult; Safety; Dose Finding; Phase 1; 3 + 3 design; Nebulizers and Vaporizers; High-Frequency Ventilation; nitric oxide; lung injury; Pulmonary Gas Exchange; Pulmonary Alveoli
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Hypoxia; Respiratory Insufficiency; Lung Injury | interventions — Nitroprusside

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nebulized sodium nitroprusside (Experimental)
  Interventions: Drug: Sodium Nitroprusside

INTERVENTIONS:
Drug: Sodium Nitroprusside — Each subject will receive one of five possible dosages of nebulized sodium nitroprusside. The dosage will be determined by the 3 + 3 dose escalation design. Only a maximum of six patients will be given a particular dosage. Arterial blood gases will be drawn at 0 min, 15 min, 30 min and 45 min during nebulized sodium nitroprusside administration. Vitals signs will be recorded every five minutes. No changes to ventilator settings or vasopressor dosage or fluid administration will be allowed.
  Other Names: Nipride, Nitropress

SUMMARY:
Acute lung injury (ALI) is caused by a wide variety of conditions, but always characterized by hypoxia and non-cardiogenic pulmonary edema. Current treatment of ALI is supportive and treatment of the underlying cause. New therapies to treat severe ALI have not been shown to improve survival, and are limited by financial and logistical resources.

The investigators propose to investigate the role of inhaled sodium nitroprusside (iSNP) in ALI. Sodium nitroprusside (SNP) is a vasodilator. When inhaled, SNP may travel to areas of the lung participating in gas exchange, and cause the blood vessels surrounding these areas to enlarge. This may result in an increase of blood vessels to these areas of the lung, and improve oxygenation. Currently, iSNP has not been studied in the adult population. Therefore, this study is intended to find the safety profile of varying doses of iSNP.

DETAILED DESCRIPTION:
Acute lung injury (ALI) is a syndrome characterized by acute hypoxemic respiratory failure with bilateral pulmonary infiltrates that are not attributed to left atrial hypertension. ALI is responsible for significant mortality and morbidity in the critically ill population.

Novel rescue therapies used to support oxygenation in severe ALI include inhaled nitric oxide and high frequency oscillatory ventilation; however, neither have been shown to reduce mortality and both are limited by logistical and financial challenges.

Inhaled sodium nitroprusside (iSNP) is a vasodilator which causes local vasodilation of pulmonary capillaries surrounding functional alveoli, resulting in improved oxygenation by redistributing pulmonary blood flow to areas with better ventilation-perfusion ratios. As iSNP can be administered by a low-cost nebulizer and is relatively inexpensive compared to other novel rescue therapies, this modality may be an alternative therapy for patients with severe hypoxemia. Two pediatric studies support the use of iSNP in ALI; however, iSNP has not been studied in the adult ALI population. To determine whether iSNP can improve oxygenation in adult ALI, the maximum tolerable dose (MTD) must first be determined.

Our study aims to determine the MTD of iSNP in adult ALI through an open-label, non-randomized, single centered, dose escalation study design, whereby subjects will receive iSNP for thirty minutes and have various physiologic variables recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Negative β-hCG in women of child bearing age (age ≤ 50)
3. Developed ALI within past 72 hours:

   * PaO2/FiO2 < 300;
   * Bilateral infiltrates on CXR;
   * No clinical evidence of elevated left atrial pressure ie. Heart failure as the cause of hypoxia and bilateral infiltrates; and
   * Recognized risk factor for ALI such as: pneumonia, aspiration pneumonitis, acute pancreatitis, massive blood transfusion, or sepsis
4. FiO2 ≥ 0.5
5. PEEP ≥ 8 cm H2O
6. Invasive arterial blood pressure line
7. Endotracheal intubation or tracheostomy
8. Conventional mechanical ventilation
9. Mean Arterial Pressure (MAP) ≥ 65 mmHg with or without use of vasopressors (stable for at least more than 1 hour)
10. Arterial pH ≥ 7.15

Exclusion Criteria:

1. Chest tube with active leak (eg. bronchopulmonary fistula),
2. Prone ventilation, inhaled nitric oxide, inhaled prostacyclin, high frequency oscillatory ventilation,
3. Lack of consent,
4. Untreated coarctation of aorta, symptomatic or severe/critical aortic stenosis as documented by echocardiogram or clinical history,
5. Evidence of increased intracranial pressure (eg. dilated pupils, known intracranial trauma or mass on head CT),
6. SpO2 <90%,
7. Contraindication to SNP i.e. hypersensitivity, congenital optic atrophy, tobacco amblyopia,
8. Active treatment with IV or transdermal nitroglycerin,
9. G6PD deficiency
10. CrCl < 30 ml/min or receiving renal replacement therapy, or
11. Total bilirubin > 68 µmol/L and AST or ALT level 2 times the upper limit of normal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerable dosage of nebulized sodium nitroprusside. This will be determined by the 3 + 3 dose finding design. | Up to 1 year
  Participants will be followed for the duration of the intervention of 45 min. . It is anticipated it will take up to 1 year to recruit the required number of participants to determine the maximum tolerable dose of nebulized sodium nitroprusside.

SECONDARY OUTCOMES:
The change in measures of oxygenation (PaO2,SaO2,oxygenation index) during iSNP administration. | 0 min, 15 min, 30 min, and 45 min
The change in heart rate (HR), mean blood pressure (MAP) during iSNP administration. | 0 min, 15 min, 30 min, and 45 min
The presence or absence of lactate, and/or methemoglobin. | 0 min, 15 min, 30 min, and 45 min

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta Mehta, MD FRCPC, Principal Investigator — Department of Critical Care Medicine, University of Toronto; Terence Ip, MD, Principal Investigator — Department of Critical Care Medicine, University of Toronto
Locations (1):
- Mount Sinai Hospital, University of Toronto, Toronto, Ontario, Canada